CLINICAL TRIAL: NCT04290936
Title: Decreasing Risk of Recurrence by TAF in HCC Patients After Curative Treatment With Low HBV Viral Load
Brief Title: Tenofovir Alafenamide(TAF) Reduces the Risk of Hepatocellular Carcinoma(HCC) Recurrence
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Yi-Hsiang Huang, M.D., Ph.D., Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IN-TW-320-5598
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: HCC Patients After Curative Treatment With Low HBV Viral Load
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Part 1: NUC-naïve patients will be randomization into tenofovir alafenamide(TAF) or placebo arm in 1:1 ratio.
  Part 2: NUCs-treated patients will be switched to tenofovir alafenamide(TAF) treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): NUC-naïve patients will be randomization into Tenofovir Alafenamide(TAF) treatment.
  Interventions: Drug: Vemlidy® (Tenofovir Alafenamide; TAF)
- Arm 2 (Placebo Comparator): NUC-naïve patients will be randomization into placebo arm.
  Interventions: Drug: Placebo
- Arm 3 (Active Comparator): NUCs-treated patients will be switched to Tenofovir Alafenamide(TAF) treatment.
  Interventions: Drug: Vemlidy® (Tenofovir Alafenamide; TAF)

INTERVENTIONS:
Drug: Vemlidy® (Tenofovir Alafenamide; TAF) — Dosage form: Oral Tablets; Dosage: 25mg; Frequency: One tablet with meals, once daily(QD).
  Arms: Arm 1; Arm 3
Drug: Placebo — Dosage form: Oral Tablets; Dosage: N/A; Frequency: One tablet with meals, once daily(QD).
  Arms: Arm 2

SUMMARY:
Hepatocellular carcinoma(HCC) is prevalent in the hepatitis B virus(HBV) infection endemic areas. For early stage of HCC, surgical resection, radiofrequency ablation (RFA) or microwave ablation (MWA) are the main treatment options. However, the risk of recurrence is as high as 50% in 5 years by surgical resection or 60-70% in 5 years by RFA. In average, the recurrence rate of HCC at 2 years is 30%. Many factors are associated with the HCC recurrence, including HBV viral load, cirrhotic stage, tumor size, tumor number, vascular invasion, alpha-fetoprotein(AFP) level and so on. Of them, high HBV viral load is associated with the risk of HCC recurrence after surgical resection, especially on late recurrence. In one previous randomized controlled trial, patients who received lamivudine, adefovir dipivoxil, or entecavir had significantly decreased early recurrence of HCC, however, whether nucleos(t)ide analogues(NUCs) can further reduce the risk of recurrence in patients with low viral loads (<2000 IU/ml) is still unclear.

In EASL 2017 guideline, all patients with compensated or decompensated cirrhosis need antiviral treatment, with any detectable HBV DNA level and regardless of alanine aminotransferase(ALT) levels. In Taiwan, even in chronic hepatitis B(CHB) infection patients with HCC, NUC is not reimbursed if their HBV viral load was less than 2000 IU/ml. It is an important unmet medical need to understanding the role of TAF in reducing the risk of recurrence in HBV-HCC patients with low HBV viral load (HBV DNA<2000 IU/ml) and significant liver fibrosis after curative treatment (The definition of significant liver fibrosis was based on reference. In our recent retrospective study, the risk of recurrence and survival are comparable between patients with and without NUCs treatment before HCC development only if NUCs treatment can be provided after curative treatment of HCC. However, a higher risk of recurrence was observed in cirrhotic patients with prior NUCs treatment before HCC occurrence. It would be interesting to investigate the incidence of recurrence by switching to tenofovir alafenamide(TAF) after curative treatment of HCC in patients already on NUCs treatment.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-positive for more than 6 months.
* HCC after curative treatment (eight by surgical resection or RFA or MWA) with significant liver fibrosis (either by Ishak≧2, Metavir≧2, Knodell≧3) or cirrhosis and HBV DNA<2,000 IU/ml.
* The duration of curative treatment of HCC to study enrollment should be less than 90 days.
* Curative treatment is confirmed by contrast-enhanced CT or MR after the surgery/RFA/MWA.

Exclusion Criteria:

* Child-Pugh class B8-C.
* Active EV bleeding within 4 weeks.
* History of hepatic encephalopathy or intractable ascites.
* BCLC C or D.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hepatocellular carcinoma(HCC) recurrence | Up to 2 years.
  Incidence of HCC recurrence

SECONDARY OUTCOMES:
Hepatocellular carcinoma(HCC) recurrence | Up to 3 years.
  HCC recurrence
Hepatocellular carcinoma(HCC) recurrence in NUCs-treated patients after switched to TAF treatment | Up to 2 years.
  HCC recurrence in NUCs-treated patients after switched to TAF treatment
Dynamic (kinetics) changes in the bio-markers related to hepatitis B virus(HBV) infection | Up to 3 years.
  HBV DNA, HBsAg, HBV RNA, HBcrAg, etc.
Changes in the renal function | Up to 3 years.
  eGFR
Changes in the bone density | Up to 3 years.
  Dual-energy X-ray absorptiometry(DEXA) scan
Regression of liver fibrosis | Up to 3 years.
  Fibroscan

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, State...
  - National Taiwan University Hospital, Taipei, State...
  - Tri-Service General Hospital, Taipei, State...
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No